CLINICAL TRIAL: NCT01698879
Title: Treatment of de Novo Acute Myeloid Leukemia With the Combination of Idarubicin, Cytarabine, and Gemtuzumab Ozogamicin (Mylotarg ®), Associated or Not Priming With G-CSF. Prospective Study of Efficacy and Toxicity
Brief Title: Prospective Study of Mylotarg and G-CSF in Acute Myeloid Leukemia Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICOG-07; 2007-006295-11 (EudraCT Number)
Record Dates: First submitted 2012-07-23; First posted 2012-10-03 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Novo Acute Myeloid Leukemia
MeSH Terms: interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm, three cohorts (Experimental): Idarubicin, cytarabine, Mylotarg.
  Interventions: Drug: Mylotarg

INTERVENTIONS:
Drug: Mylotarg — Cohort 1 version 1.0. GO: 6mg/m^2 (maximum 10 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine: 100 mg/m^2 IV days 1 to 7, to begin 4 hours after the administration of GO.
  Cohort 1.0 version 2.0: GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine: 100 mg/m^2 IV days 1 to 7, to begin 4 hours after the administration of GO.
  Cohort 2: G-CSF: 150 mcg/m^2, SC, days 0 to 7. GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine: 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours later after the administration of GO.

SUMMARY:
Acute myeloid leukemia (AML) is a neoplasm of immature hematopoietic cells (blasts) with altered ripening capacity. Due to excessive proliferation, the blasts displace normal hematopoietic cells and bone marrow failure appears. Leukemic cells also infiltrate extramedullary tissues.

Following the standard chemotherapy treatment, the CR rate achieved is around 65-75% for all patients and 15% lower when considering only patients over 65 years. Modifications to the standard regimen consist of replacing the DNR for a cytotoxic one, modifying the dose of ara-C or adding a third drug.

Gemtuzumab ozogamicin (Mylotarg ®) is an immunoconjugate between anti-CD33 antibody and a cytotoxic antitumor antibiotic, calicheamicin. Mylotarg ® antibody specifically binds to CD33, a sialic acid-dependent adhesion protein expressed in over 90% of LMA10. Mylotarg ® selectively transports the cytotoxic agent calicheamicin into leukemic cells and hematopoietic progenitors differentiated from the myelomonocytic line, while respecting the pluripotent hematopoietic stem cells. Calicheamicin is released only after the fixation of the antibody anti-CD33 and its internalization by the cell, after which binds to and damages the DNA.

Mylotarg ® is approved in the U.S. for the treatment of CD33 positive AML in first relapse, for patients older than 60 years non-candidates for other intensive treatment modalities.

Since the efficacy of Mylotarg ® is equivalent and its toxicity profile less than the conventional therapy, it is logical to conduct a phase II trial exploring the role of Mylotarg ® in the early stages of treatment of AML.

Previous experience with gemtuzumab ozogamicin in relapsed patients led to its use combined with induction chemotherapy. The aim was to improve the CR rate reached with the latter and reduce relapse after achieving greater leukemic cytoreduction.

Recent data from the HOVON group support that the administration of G-CSF before and during induction chemotherapy decreases the incidence of relapse in patients with AML, particularly those considered to have intermediate risk.

Everything mentioned above justifies to investigate the combination of GO combined with chemotherapy with IDR and ara-C in standard 3x7 scheme and analyze the effect of sensitization with G-CSF in patients with AML de novo. If the treatment proposed here is effective and presents an acceptable toxicity it should be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary or "de novo" AML, different than promyelocytic or M3 subtype.
2. Age 18 to 70 years.
3. Written informed consent form

Exclusion Criteria:

1. Acute leukemia appeared after a myeloproliferative process or a myelodysplastic syndrome longer than 6 months, AML arising after another cured malignant disease (e.g. Hodgkin's disease), and secondary AML treated with alkylating agents or radiation.
2. Acute promyelocytic leukemia.
3. Relevant history of liver disease. Significant impaired liver function (bilirubin, AST or ALT ≥ 2.5 times the normal value) not attributable to leukemic infiltration.
4. Patients with prior heart failure.
5. Symptomatic chronic respiratory failure.
6. Positive serology for HIV, hepatitis C virus or its surface antigen.
7. Estimated life expectancy less than 3 months, despite treatment.
8. Pregnancy or breastfeeding at the time of inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-10; Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Sierra, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (6):
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Version 1.0: Mylotarg: Cohort 1 version 1.0 (5 evaluable patients):
  GO: 6 mg/m^2 (maximum 10 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
  If chemo-sensitivity is observed after a first course of treatment (50% or more reduction of blasts compared to baseline) a second identical cycle will be administered.
- Cohort 1 Version 2.0: Idarubicin, cytarabine, Mylotarg
  Mylotarg: Cohort 1 (20 evaluable patients):
  GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
- Cohort 2: Cohort 2 (20 evaluable patients):
  G-CSF: 150 mcg/m^2, SC, days 0 to 7, to begin 12 to 18 hours before treatment with Gemtuzumab. GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1.
  Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours later after the administration of GO.
Period: Overall Study
Arm/Group | Cohort 1 Version 1.0 | Cohort 1 Version 2.0 | Cohort 2
Started | 6 | 20 | 20
Completed | 5 | 20 | 20
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: From cohort 1 version 1.0, one patient did not receive any study treatment (PIS withdrawal), for that reason is not considered for outcome assessment.
Groups:
- Cohort 1, Version 1.0: Mylotarg: Cohort 1 version 1.0 (5 evaluable patients):
  GO: 6 mg/m^2 (maximum 10 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
  If chemo-sensitivity is observed after a first course of treatment (50% or more reduction of blasts compared to baseline) a second identical cycle will be administered.
- Cohort 1, Version 2.0: Mylotarg: Cohort 1 (20 evaluable patients):
  GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4.
  Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Version 1.0 | Cohort 1, Version 2.0 | Cohort 2 | Total
Number analyzed (Participants) | 5 | 20 | 20 | 45
Age, Continuous [Median (Full Range); unit: years] | 56 [32 to 61] | 49 [22 to 64] | 61 [24 to 69] | 61 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The first 5 patients received GO 6mg/m2 but this dose was halted by unacceptable toxicity. Therefore, in Cohort 1 were included 20 patients receiving IA plus 3 mg/m2 GO. Cohort 2 included 20 patients who received treatment as in cohort 1 plus G-CSF priming
  Participants
    Female | 2 | 9 | 5 | 16
    Male | 3 | 11 | 15 | 29
Region of Enrollment [Number; unit: participants] — Population: One patient has not been evaluated because has not received study treatment.
  participants
    Spain | 5 | 20 | 20 | 45
Leucocites at diagnosis [Median (Full Range); unit: Cells x 10^9/L] — Population: The first 5 patients received GO 6mg/m2 but this dose was halted by unacceptable toxicity. Therefore, in Cohort 1 were included 20 patients receiving IA plus 3 mg/m2 GO. Cohort 2 included 20 patients who received treatment as in cohort 1 plus G-CSF priming.
  Cells x 10^9/L | 13.48 [2.1 to 31.85] | 7.66 [1 to 96.6] | 6.96 [0.9 to 114] | 6.96 [0.9 to 114]
Citogenetic [Count of Participants; unit: Participants] — Population: 1 patient not evaluable because has not received study treatment.
  Participants
    Favorable | 1 | 5 | 3 | 9
    Intermediate | 3 | 13 | 12 | 28
    Adverse | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission of the Disease
Description: Rate of patients that have obtained complete remission. Complete remission is defined as, bone marrow normocellular or slightly hypocellular with proportion of blasts <5%, including the erythroid cell count (and including promonocytes in case of M5), no Auer rods, no extramedullary leukemia, neutrophils and platelets rising. The persistence of minimal residual disease in immunophenotypic study will not invalidate the standard cytogenetic complete remission.
Time Frame: 28 days after chemotherapy
Population: Initial 5 patients included in cohort 1 version 1.0 (closed due toxicity) have been evaluated for safety outcome but not evaluated for efficacy because the treatment is not feasible.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Version 1.0 | Cohort 1, Version 2.0 | Cohort 2
Number analyzed (Participants) | 5 | 20 | 20
Participants
  Complete Response | NA — It has not been evaluated efficacy result of this cohort with unacceptable toxicity profile | 18 | 16
  Partial Response | NA — It has not been evaluated efficacy result of this cohort with unacceptable toxicity profile | 1 | 2
  Refractory | NA — It has not been evaluated efficacy result of this cohort with unacceptable toxicity profile | 1 | 2

2. Secondary Outcome: Secondary Toxicity to Mylotarg(R)
Description: Hematological toxicity, hepatic and gastrointestinal toxicity, fever and infections, pulmonary complications, duration of hospitalization
Time Frame: Baseline, weekly during treatment and at month 3 and month 6 after first induction.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1, Version 1.0: Initial 5 patients of cohort 1 (closed due toxicity)
- Cohort 1, Version 2.0: Idarubicin, cytarabine, Mylotarg
  Mylotarg: Cohort 1 (20 evaluable patients):
  GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
Arm/Group | Cohort 1, Version 1.0 | Cohort 1, Version 2.0 | Cohort 2
Number analyzed (Participants) | 5 | 20 | 20
percentage of participants
  Grade IV Hematologic toxicity | 0 | 100 | 95
  Grade II Hematologic toxicity | 0 | 0 | 5
  Grade I/II Hepatic toxicity | 20 | 10 | 10
  Grade III/IV hepatic toxicity | 40 | 5 | 15
  Grade I/II Infection | 0 | 10 | 25
  Grade III/IV Infection | 0 | 5 | 30

3. Secondary Outcome: Mortality at Induction
Description: all deaths occurring after the first administration of MylotargTM until the time of transplantation with no leukemic relapse has occurred, and all deaths in the 6 first months after administration of the second dose of MylotargTM with no leukemic relapse occurred.
Time Frame: Weekly during treatment, at third month and at 6 months after last administration of Mylotarg
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Version 2.0: Mylotarg: Cohort 1 (20 evaluable patients):
  GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
Arm/Group | Cohort 1, Version 1.0 | Cohort 1 Version 2.0 | Cohort 2
Number analyzed (Participants) | 5 | 20 | 20
Participants | 1 | 0 | 2

4. Secondary Outcome: Capacity to Obtain Hematopoietic Progenitor Cells (HPC) for Autotransplantation - DATA NOT COLLECTED
Description: Rate of patients with capacity to obtain hematopoietic progenitor cells (HPC) for autotransplantation. This analysis has not been performed, because data were not available in sites.
Time Frame: One month before transplant, expected at 9 months after end of treatment.
Population: Initial 5 patients included in cohort 1 version 1.0 (closed due toxicity) have been evaluated for safety outcome but not evaluated for efficacy because the treatment is not feasible. This analysis has not been performed because data were not available for any of the cohorts studied.
Arm/Group | Cohort 1, Version 1.0 | Cohort 1, Version 2.0 | Cohort 2
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Relapse After 6 Months
Description: Rate of patients that have relapse after 6 months of obtained complete remission.
Time Frame: 6 months from complete remission
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1, Version 2.0: Idarubicin, cytarabine, Mylotarg.
  Mylotarg: Cohort 1 (20 evaluable patients):
  GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
Arm/Group | Cohort 1, Version 2.0 | Cohort 2
Number analyzed (Participants) | 20 | 20
percentage of participants | 30 | 59

6. Secondary Outcome: Survival After 6 Months
Description: rate of patients alive within 6 months of obtained complete remission
Time Frame: 6 months after complete remission
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1: Idarubicin, cytarabine, Mylotarg, G-CSF.
  Mylotarg: Cohort 1 (20 evaluable patients):
  GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1. Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 20 | 20
percentage of participants | 80 | 80

ADVERSE EVENTS:
Time Frame: From October 2008 up to September 2016, 7 years and 11 months.
Groups:
- 5 Patients Treated in Trial With Prrotocol Version 1.0: Idarubicin, cytarabine, Mylotarg, G-CSF.
  Mylotarg::
  GO: 5 mg/m^2 (maximum 10 mg), IV infusion, 2 hours, day 1. If no adequate response, GO: 3 mg/m^2 (maximum 5 mg), IV infusion, 2 hours, day 1.
  Idarubicin: 12 mg/m^2, IV, 30 minutes, on days 2, 3, 4. Cytarabine (cytosine arabinoside): 100 mg/m^2 IV continuous infusion on days 1 to 7, to begin 4 hours after the administration of GO.
Arm/Group | Cohort 1 | Cohort 2 | 5 Patients Treated in Trial With Prrotocol Version 1.0
All-Cause Mortality (participants affected / at risk) | 1/20 | 2/20 | 1/5
Serious Adverse Events (participants affected / at risk) | 3/20 | 6/20 | 2/5
Other Adverse Events (participants affected / at risk) | 20/20 | 19/20 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=20) | Cohort 2 (N=20) | 5 Patients Treated in Trial With Prrotocol Version 1.0 (N=5)
Transient Ischemic event (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Severe respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Toxic megacolon (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Liver failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Toxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=20) | Cohort 2 (N=20) | 5 Patients Treated in Trial With Prrotocol Version 1.0 (N=5)
Grade 4 hematologic toxicity (Blood and lymphatic system disorders) | 20 (20) | 19 (19) | 3 (3)
G1/2 Hepatic toxicity (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0)
G3/G4 Hepatic Toxicity (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0)
Grade I/II infectous toxicity (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Grade 3 Infectous toxicity (Infections and infestations) | 1 (1) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days